CLINICAL TRIAL: NCT01550042
Title: Extended Rhythm SCreening for AtRial Fibrillation in Cryptogenic Stroke Patients
Acronym: SCARF
Status: Terminated | Type: Observational
Why Stopped: Inclusion rate problems, not enough eligible patients
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, B. Oude Velthuis, Research fellow electrophysiology, Medisch Spectrum Twente
Other Study IDs: NL36491.044.11; P11-25 (Other: METC Twente)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intensive observation cohort: Patients > 18 years of age diagnosed with a recent episode of cryptogenic stroke with long term rhythm observation using an implantable loop recorder for detecting atrial fibrillation.

SUMMARY:
Recent studies demonstrated that prolonged rhythm observation increases the detection of atrial fibrillation in patients prior diagnosed as cryptogenic stroke. Detection of atrial fibrillation in these patients has important therapeutic implications for the anticoagulation regimen. However, data on optimal monitoring duration and method of AF detection are limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age Recent episode (≤60 days) of cryptogenic ischemic stroke
* Undetermined etiology with negative evaluation (including cardioembolism work- up) according to the criteria for the Trial of Org 10172 in Acute Stroke Treatment (TOAST)
* Implantation of an implantable loop recorder within two months after index event
* Able of providing informed consent

Exclusion Criteria:

* Pre-existing indication for vitamin K antagonist
* Untreated hyperthyroidism
* Indication for pacemaker implantation, implantable cardioverter defibrillator (ICD) or Cardiac Resynchronisation Therapy (CRT)
* Severe co-morbidity not likely to complete follow-up for one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with a ischemic stroke of undetermined etiology
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Documented Atrial Fibrillation (AF) | One year
  The percentage of patients with documented AF based on implantable cardiac monitor registration during a follow-up period of at least 12 months after an episode of cryptogenic stroke.

SECONDARY OUTCOMES:
Time to documented AF | One year
  Time to documented AF using an Implantable Loop Recorder (ILR) data
Recurrent stroke | One year
  Incidence of recurrent stroke

CONTACTS AND LOCATIONS:
Overall Officials: Marcoen Scholten, MD PhD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente / Thoraxcenter, Enschede, Overijssel, Netherlands

REFERENCES:
- See also: Thoraxcenter — http://www.mst.nl/thoraxcentre/